CLINICAL TRIAL: NCT07288840
Title: Exercise Prescription in Cardiac Rehabilitation Mediated by Autonomic Function
Acronym: EXCARMA
Status: Enrolling by invitation | Type: Observational
Sponsor: Instituto Politécnico de Leiria (Other)
Collaborators: Universidade do Minho - ICVS (Unknown); Hospital Santo André - Centro Hospitalar de Leiria (Unknown); Fundação para a Ciência e a Tecnologia (FCT) (Unknown)
Responsible Party: Principal Investigator, Alexandre Antunes, Medical Doctor (MD), Cardiologist, Coordinator of the Cardiac Rehabilitation Unit of Hospital Santo André, Instituto Politécnico de Leiria
Other Study IDs: FCT 2024.04320.BD
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Rehabilitation; Exercise Therapy; Autonomic Nervous System Imbalance; Treatment Outcomes
Keywords: Cardiac Rehabilitation; Exercise prescription; Autonomic funtion; microneurography; cardiopulmonary exercise testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for serum catecholamine measurement and urine samples for urinary catecholamine analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Coronary artery disease without Heart Failure (CADnonHF): This group with clearly demonstrated Autonomic Simpathetic System overactivation will have a detailed evaluation of the autonomic nervous system by performing an echocardiogram, 24-hour Holter monitoring, cardiopulmonary exercise test, long-term electrocardiogram, microneurography, and serum and urinary determination of catecholamine levels
- Patients with non- ischemic Heart Failure with reduced ejection fraction (NIHFrEF): This group, that also has clearly demonstrated Autonomic Simpathetic System overactivation, will, in the same way, have a detailed evaluation of the autonomic nervous system by performing an echocardiogram, 24-hour Holter monitoring, cardiopulmonary exercise test, long-term electrocardiogram, microneurography, and serum and urinary determination of catecholamine levels

SUMMARY:
Cardiac rehabilitation (CR) is an essential secondary prevention component in the treatment of cardiovascular diseases and one of the most cost- effective clinical interventions. Exercise training (ET) in CR programs (CRP) has unequivocal benefits in the reduction of cardiovascular adverse events, by decreasing the overactivated sympathetic tone. This ET added value can be measured by variables that express autonomic control using indirect (standard) or direct (experimental) methodologies. Direct autonomic assessment (ex. Microneurography) is accurate but unusable in daily practice, whereas standard indirect autonomic assessment using clinical parameters is imprecise, resulting in underprescription to safeguard patient safety, with less benefit to the patients. In this project, we aim to apply Machine Learning models to a set of indirect and direct variables, to make a multivariate correlation analysis and so define a normalization factor for exercise prescription.

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) has proved to be an essential secondary prevention component of the continuum in the treatment of Cardiovascular diseases (CVD), being a Class I recommendation with level of evidence A and B on the European Society of Cardiology (ESC) and American Heart Association and American College of Cardiology (AHA/ACC) Guidelines. CR is also one of the most cost-effective clinical interventions in the treatment of CVD. These diseases, namely coronary artery disease (CAD) and heart failure (HF), are associated with autonomic dysfunction, particularly an overactivation of the autonomic sympathetic system (ASS), leading to coronary vasoconstriction, myocardial remodeling, and increased basal oxygen consumption. The main component of the CR programs (CRP) is Exercise training (ET), one of the central pillars of non- pharmacological treatment in CVD, thus preventing the above- mentioned progression of deleterious effects. The role of ET in CRP has been increasingly emphasized; however, it is still not clear, among the variety of existing training programs, which is the optimal combination and type of exercise (aerobic/anaerobic or both), frequency and duration of the sessions, whose prescription should be customized considering the patient's clinical history and the pre-CRP exam results. This limitation is pointed out as a major drawback in obtaining optimized results on CRP. The absence of a methodology that can more precisely assess and hence better quantify the effect of the prescription, safely optimizing the training plan, is one of the central problems regarding CR, and will be addressed in this research proposal putting the autonomic modulation of CV system in the center of the rational to prescribe ET in CRP. The main objective of this research plan is to draw an objective and individualized protocol to prescribe ET in CRPs based on the Autonomic output.

After careful ponderation, two important but different pathologies with clearly demonstrated ASS overactivation were considered: "non- ischemic HF with reduced ejection fraction" (NIHFrEF) and "CAD without HF" (CADnonHF). The following secondary objectives contribute to the achievement of this central goal, and define the majority of the associated tasks:

* Evaluation of the basal sympathetic activation pattern in patients with NIHFrEF and CADnonHF (Task2);
* Definition of a normalization factor regarding sympathetic activation for ET prescription purposes in the context of CRPs (Task3)
* Definition of an exercise training program for CRPs with prescription guided by the autonomic response (Task 4); In Task 2 the basal activation level of the Autonomic nervous system (ANS) will be characterized for each of the two identified conditions (NIHFrEF and CADnonHF) using a sample of 30 patients for each one to ensure a good approximation of the sampling distribution of the mean using the central limit theorem, and the participants will be enrolled at the CR consultation in Centro Hospitalar de Leiria (CHL) Cardiology department. The CHL CR Unit is accreditated by the European Association of Preventive Cardiology (EAPC) since 2022. Classical indirect measures of ANS which are relatively imprecise, such as heart rate variability (HRV) and derived indexes will be obtained with a 24h Holter and a "long duration EKG", as well as the first minute HR recovery with a Cardiopulmonary Exercise Test (CPET) and also serum catecholamines in blood and urine samples. Besides these indirect measures, a direct recording of the SNS obtained by microneurography (MSNA) will be conducted, being available at the host research institution (ciTechCare). The set of variables (autonomic and its derivatives), together with the metabolic biomarkers, will allow a multivariate correlation analysis followed by the use of the Machine Learning algorithm "Principal Component analysis" (PCA) to reduce the dimensionality of the data set, and so define a normalization factor for exercise prescription purposes, which corresponds to the main goal associated with Task 3. This normalization factor will be key to establish the individual pattern of sympathetic activation, establishing the same starting point for initial prescription of exercise and an unbiased follow up of patient's performance. Regarding Task 4, training plans (aerobic/anaerobic load) will be carried out in conjunction with the levels defined for the classification model (one of the derivable of the previous Task), and will be developed by the candidate along with the Physiatrist of the CRP Team, by setting a combined (aerobic and resistance) and stratified (with various levels of intensity, frequency, stages and duration) training program. This protocol will be evaluated by the due health ethics committees (Task 1), and all legal issues regarding safety and data protection will be respected.

Regarding risks and strategies to mitigate them, the main risk is related to data assessment. In that case other hospitals may be contacted to increase the number of participants. Another risk is related to task dependency. In this case, the experience of the mentors and the integration of this project in a team with expertise in CRP and familiar with artificial intelligence applications in Medicine will be determinant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Coronary artery disease and no heart failure criteria
* Patients with non ischaemic heart failure and reduced left ventricle ejection fraction

Exclusion Criteria:

* patients with ongoing acute coronary syndrome
* patients with ongoing acute decompensated heart failure
* Severe valvular heart disease that might confound the relationship between exercise and autonomic function.
* Severe arrhythmias (e.g., sustained ventricular tachycardia, atrial fibrillation with a rapid ventricular rate) that are symptomatic or untreated
* Severe uncontrolled hypertension (e.g., systolic BP > 180 mmHg or diastolic BP > 110 mmHg)
* Active infectious diseases or other significant acute medical illnesses (e.g., sepsis, active malignancy, acute kidney injury)
* Pregnancy or lactation (to ensure safety during exercise interventions)
* Significant cognitive impairment or mental illness (e.g., dementia, schizophrenia) that would impair the ability to follow exercise protocols or understand study instructions
* nability to comply with study procedures due to any reason (e.g., language barriers, lack of informed consent)
* Chronically immunocompromised states (e.g., HIV with CD4 count < 200 cells/µL or on immunosuppressive therapy)
* Presence of significant comorbidities such as advanced chronic obstructive pulmonary disease (COPD), kidney disease (e.g., stage 4-5 chronic kidney disease), or uncontrolled diabetes that would make exercise unsafe or confound the study outcomes
* Critical limb ischemia, or severely symptomatic peripheral artery disease or claudication limiting functional capacity and response to exercise
* Advanced chronic kidney disease (stage 4 or 5), due to contraindications with exercise
* Severe anemia (hemoglobin < 8 g/dL) or other blood disorders that affect exercise capacity
* Inability to tolerate exercise due to other comorbidities or debility
* individuals with known autonomic neuropathy (such as poorly controlled diabetes or neurodegenerative disorders)

Specific Exclusion Criteria for Coronary Artery Disease (CAD) without Heart Failure Group:

* Left ventricular ejection fraction (LVEF) < 50%
* Clinical/echocardiographic criteria of heart failure with oreserved ejection fraction.

Specific Exclusion Criteria for Non-Ischemic Heart Failure with Reduced LVEF Group:

* Ischemic heart disease or previous myocardial infarction
* LVEF > 40%
* End-stage heart failure (e.g., patients on a heart transplant list, those with imminent need for mechanical circulatory support like LVAD).
* Severe fluid overload that cannot be corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with non-ischemic heart failure with reduced ejection fraction (NIHFrEF) or stable coronary artery disease without heart failure (CADnonHF), consecutively enrolled in the Cardiac Rehabilitation Program at Centro Hospitalar de Leiria, and undergoing comprehensive autonomic and metabolic assessment."
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Normalization Factor for Sympathetic Activation Derived from Multimodal Autonomic Assessment | Baseline (before initiation of cardiac rehabilitation program)
  A composite autonomic normalization factor will be generated using Principal Component Analysis (PCA) applied to multimodal autonomic and metabolic biomarkers (including microneurography-derived MSNA, heart rate variability indices from 24-hour Holter, CPET first-minute heart rate recovery, and serum/urinary catecholamines). This factor will quantify the individual degree of sympathetic activation and will serve as the basis for personalized exercise training prescription (Units of mesaure: unitless)

SECONDARY OUTCOMES:
Basal Sympathetic Nervous System Activity (MSNA burst frequency) | Baseline
  Direct sympathetic activity will be quantified using microneurography (sympathetic nerve activity, MSNA), expressed as bursts/minute (bursts/min), to characterize autonomic dysfunction in NIHFrEF and CADnonHF groups.
SDNN (Heart Rate Variability) obtained from 24-hour Holter ECG and long-duration ECG | Baseline
  Standard deviation of normal-to-normal intervals as an index of overall HRV (Unit of Measure: milliseconds - ms)
RMSSD (Heart Rate Variability) obtained from 24-hour Holter ECG and long duration ECG | Baseline
  Root mean square of successive differences as a measure of parasympathetic activity (Unit of Measure: ms²)
LF Power (Heart Rate Variability) Low-frequency spectral power obtained from 24-hour Holter ECG | Baseline
  LF component of HRV as an index of sympathetic/parasympathetic modulation (Units ms²)
LF/HF Ratio (Heart Rate Variability) obtained from 24-hour Holter ECG | Baseline
  Ratio of low-frequency to high-frequency power reflecting autonomic balance (Unit of Measure: unitless)
Plasma epinephrine concentration | Baseline
  Quantified by blood sample to assess biochemical sympathetic activity. Unit of Measure: pg/mL
Plasma norepinephrine concentration | Baseline
  Quantified by blood sample to assess sympathetic activation (Unit of Measure: pg/mL)
Plasma dopamine concentration | Baseline
  Quantified by blood sample to assess catecholaminergic activity (units of measure pg/mL)
Urinary metanephrine | Baseline
  24-hour urinary excretion as an index of catecholamine metabolism (unit of measure µg/24h)
Urinary normetanephrine | Baseline
  24-hour urinary excretion measurement (unit of measure: µg/24h)
Urinary 3-methoxytyramine | Baseline
  24-hour urinary excretion measurement (unit of measure - µg/24h)
CPET First-Minute Heart Rate Recovery | Baseline
  Difference between peak HR and HR at 1-minute post-exercise during cardiopulmonary exercise test, reflecting parasympathetic reactivation (units of measure: beats per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Vitor Hugo Eira Pereira, MD, PhD, Study Director — ICVS - Life and Health Sciences Research Institute, Minho University Medical School; Rui Manuel Fonseca Pinto, MD, PhD, Study Director — ciTechCare - Center for Innovative Care and Health Technology, Polytechnic University of Leiria; João Carlos Araújo Morais, MD,PhD, Study Director — ciTechCare - Center for Innovative Care and Health Technology
Locations (2):
- Portugal (2):
  - ciTechCare - Center for Innovative Care and Health Technology, Leiria, Leiria District
  - ICVS - Life and Health Sciences Research Institute, Minho University Medical School, Braga, Minho

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study collects sensitive physiological and clinical information that carries a high risk of re-identification, and current institutional and regulatory constraints do not permit external data sharing.

REFERENCES:
- [Background] Anderson L, Thompson DR, Oldridge N, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2016 Jan 5;2016(1):CD001800. doi: 10.1002/14651858.CD001800.pub3. PMID 26730878
- [Background] Watson AM, Hood SG, May CN. Mechanisms of sympathetic activation in heart failure. Clin Exp Pharmacol Physiol. 2006 Dec;33(12):1269-74. doi: 10.1111/j.1440-1681.2006.04523.x. PMID 17184514
- [Background] Townsend N, Wilson L, Bhatnagar P, Wickramasinghe K, Rayner M, Nichols M. Cardiovascular disease in Europe: epidemiological update 2016. Eur Heart J. 2016 Nov 7;37(42):3232-3245. doi: 10.1093/eurheartj/ehw334. Epub 2016 Aug 14. No abstract available. PMID 27523477
- [Background] Bento L, Fonseca-Pinto R, Povoa P. Autonomic nervous system monitoring in intensive care as a prognostic tool. Systematic review. Rev Bras Ter Intensiva. 2017 Oct-Dec;29(4):481-489. doi: 10.5935/0103-507X.20170072. PMID 29340538
- [Background] Sacramento JF, Ribeiro MJ, Rodrigues T, Olea E, Melo BF, Guarino MP, Fonseca-Pinto R, Ferreira CR, Coelho J, Obeso A, Seica R, Matafome P, Conde SV. Functional abolition of carotid body activity restores insulin action and glucose homeostasis in rats: key roles for visceral adipose tissue and the liver. Diabetologia. 2017 Jan;60(1):158-168. doi: 10.1007/s00125-016-4133-y. Epub 2016 Oct 16. PMID 27744526
- [Background] Sandesara PB, Lambert CT, Gordon NF, Fletcher GF, Franklin BA, Wenger NK, Sperling L. Cardiac rehabilitation and risk reduction: time to "rebrand and reinvigorate". J Am Coll Cardiol. 2015 Feb 3;65(4):389-395. doi: 10.1016/j.jacc.2014.10.059. PMID 25634839
- [Background] Adler AJ, Martin N, Mariani J, Tajer CD, Owolabi OO, Free C, Serrano NC, Casas JP, Perel P. Mobile phone text messaging to improve medication adherence in secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2017 Apr 29;4(4):CD011851. doi: 10.1002/14651858.CD011851.pub2. PMID 28455948
- [Background] Besnier F, Labrunee M, Pathak A, Pavy-Le Traon A, Gales C, Senard JM, Guiraud T. Exercise training-induced modification in autonomic nervous system: An update for cardiac patients. Ann Phys Rehabil Med. 2017 Jan;60(1):27-35. doi: 10.1016/j.rehab.2016.07.002. Epub 2016 Aug 16. PMID 27542313
- [Background] Long L, Anderson L, He J, Gandhi M, Dewhirst A, Bridges C, Taylor R. Exercise-based cardiac rehabilitation for stable angina: systematic review and meta-analysis. Open Heart. 2019 Jun 5;6(1):e000989. doi: 10.1136/openhrt-2018-000989. eCollection 2019. PMID 31245012
- [Background] Alter DA, Zagorski B, Marzolini S, Forhan M, Oh PI. On-site programmatic attendance to cardiac rehabilitation and the healthy-adherer effect. Eur J Prev Cardiol. 2015 Oct;22(10):1232-46. doi: 10.1177/2047487314544084. Epub 2014 Jul 30. PMID 25079239
- [Background] Andrade N, Alves E, Costa AR, Moura-Ferreira P, Azevedo A, Lunet N. Knowledge about cardiovascular disease in Portugal. Rev Port Cardiol (Engl Ed). 2018 Aug;37(8):669-677. doi: 10.1016/j.repc.2017.10.017. Epub 2018 Jul 25. English, Portuguese. PMID 30055948
- [Background] Abreu A, Mendes M, Dores H, Silveira C, Fontes P, Teixeira M, Santa Clara H, Morais J. Mandatory criteria for cardiac rehabilitation programs: 2018 guidelines from the Portuguese Society of Cardiology. Rev Port Cardiol (Engl Ed). 2018 May;37(5):363-373. doi: 10.1016/j.repc.2018.02.006. Epub 2018 Apr 30. English, Portuguese. PMID 29724635
- [Background] Atlas Writing Group; ESC Atlas of Cardiology is a compendium of cardiovascular statistics compiled by the European Heart Agency, a department of the European Society of Cardiology.; Developed in collaboration with the national societies of the European Society of Cardiology member countries; Timmis A, Townsend N, Gale CP, Torbica A, Lettino M, Petersen SE, Mossialos EA, Maggioni AP, Kazakiewicz D, May HT, De Smedt D, Flather M, Zuhlke L, Beltrame JF, Huculeci R, Tavazzi L, Hindricks G, Bax J, Casadei B, Achenbach S, Wright L, Vardas P. European Society of Cardiology: Cardiovascular Disease Statistics 2019 (Executive Summary). Eur Heart J Qual Care Clin Outcomes. 2020 Jan 1;6(1):7-9. doi: 10.1093/ehjqcco/qcz065. No abstract available. PMID 31957796